CLINICAL TRIAL: NCT01406769
Title: A Limited Access Phase II Trial Utilizing Bioimpedance to Measure Lower Extremity Lymphedema Associated With the Surgical Management of a Vulvar Cancer
Brief Title: Bioimpedance Spectroscopy in Detecting Lower-Extremity Lymphedema in Patients With Stage I, Stage II, Stage III, or Stage IV Vulvar Cancer Undergoing Surgery and Lymphadenectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GOG-0269; NCI-2011-03798 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000706551; GOG-0269 (Other: Gynecologic Oncology Group); GOG-0269 (Other: DCP); GOG-0269 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Lymphedema; Perioperative/Postoperative Complications; Stage IA Vulvar Cancer AJCC v7; Stage IB Vulvar Cancer AJCC v7; Stage II Vulvar Cancer AJCC v7; Stage IIIA Vulvar Cancer AJCC v7; Stage IIIB Vulvar Cancer AJCC v7; Stage IIIC Vulvar Cancer AJCC v7; Stage IVA Vulvar Cancer AJCC v7; Stage IVB Vulvar Cancer AJCC v6 and v7
MeSH Terms: conditions — Lymphedema; Postoperative Complications; Vulvar Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (bioimpedance to measure lymphedema) (Experimental): Patients undergo preoperative and postoperative lower-extremity lymphedema assessment comprising serial circumferential measurements, bioimpedance spectroscopy measurements, and clinical evaluation using the Stemmer sign. Patients undergo radical vulvectomy or radical local excision as prescribed by GOG-0244, and unilateral or bilateral inguinal or inguinal-femoral lymphadenectomy.
  Interventions: Procedure: Bioelectric Impedance Analysis; Procedure: Lymphadenectomy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Bioelectric Impedance Analysis — Undergo preoperative and postoperative lower-extremity lymphedema assessment
  Other Names: BIA; Bioelectric Impedance; Bioelectric Impedance Test; Bioelectrical Impedance Analysis; Bioimpedance Analysis
Procedure: Lymphadenectomy — Undergo lymphadenectomy
  Other Names: excision of the lymph node; Lymph Node Dissection; lymph node excision
Procedure: Therapeutic Conventional Surgery — Undergo radical vulvectomy or radical local excision

SUMMARY:
This phase II trial studies bioimpedance spectroscopy in detecting lower-extremity lymphedema in patients with stage I, stage II, stage III, or stage IV vulvar cancer undergoing surgery and lymphadenectomy. Diagnostic procedures, such as bioimpedance spectroscopy, may help doctors to predict the onset of lower-extremity lymphedema in patients with vulvar cancer undergoing surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To evaluate the sensitivity, specificity, and feasibility of bioimpedance technology as compared to clinically derived measurements to include circumferential volumetric measurements to detect lower-extremity lymphedema in patients who are undergoing an inguinal lymphadenectomy during the concurrent surgical management of a vulvar cancer.

OUTLINE: This is a multicenter study.

Patients undergo preoperative and postoperative lower-extremity lymphedema assessment comprising serial circumferential measurements, bioimpedance spectroscopy measurements, and clinical evaluation using the Stemmer sign. Patients undergo radical vulvectomy or radical local excision as prescribed by GOG-0244, and unilateral or bilateral inguinal or inguinal-femoral lymphadenectomy.

After completion of study, patients are followed up at 4-6 weeks, every 3 months for 1 year, and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vulvar cancer already enrolled onto Gynecologic Oncology Group (GOG)-0244 who will undergo or have undergone definitive surgery for primary stage I-IV vulvar cancer who will receive a radical vulvectomy or radical local excision with concurrent unilateral or bilateral inguinal or inguinal-femoral lymphadenectomy;

  * Patients who are going to receive multi-modality therapy (radiation +/- chemotherapy) after undergoing surgery are eligible
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information for GOG-0269 and for GOG-0244
* Patients may undergo sentinel node mapping as long as it is followed by a full lymphadenectomy during the same operative event
* Serum Albumin level of >= 3.0 within 14 days of entry
* Patients with a GOG performance status of 0, 1, or 2

Exclusion Criteria:

* Patients not enrolled onto GOG-0244
* Patients with any prior clinical history of lower extremity lymphedema
* Patients who have a history of congestive heart failure, chronic renal disease, or chronic liver disease
* Patients with a prior history of chronic lower extremity swelling
* Patients with a GOG Performance Grade of 3 or 4
* Patients with a history of other invasive malignancies if that malignancy included a bilateral lymph node procedure (example: bilateral mastectomies and axillary lymphadenectomies) or if their previous cancer treatment included any of the surgical procedures
* Patients who have had prior lower extremity vascular surgery (arterial or venous)
* Patients who have had prior pelvic bilateral axillary or any pelvic, abdominal, inguinal, or lower extremity radiation therapy
* Patients who are going to receive another elective surgery during the same operative event as their inguinal lymphadenectomy and vulvar surgery
* Patients who undergo sentinel node biopsy without the intention of undergoing a complete lymphadenectomy during that same operative event
* Patients with an implanted cardiac device such as a pacemaker or implantable cardioverter defibrillator
* Patients who are pregnant or currently breastfeeding
* Patients who have been treated for, or are at risk of, bilateral arm lymphedema
* Patients with an allergic reaction to electrocardiogram (EKG) electrodes
* Patients who have had bilateral auxiliary dissection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-07-16 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity, and feasibility of bioimpedance technology as compared to clinically derived measurements (limb volume and Stemmer Sign) | Up to 24 months post-operatively
  The usual assessment of sensitivity and specificity using the volume based diagnosis as the ?Gold Standard? after an receiver operating characteristic (ROC) analysis to determine the cut-point for the definition of a diagnosis of lymphedema by the bioimpedance method will be performed.
Frequency and severity of adverse events using Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jay W Carlson, Principal Investigator — Gynecologic Oncology Group
Locations (11):
- United States (11):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mercy Hospital Springfield, Springfield, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin